CLINICAL TRIAL: NCT01938040
Title: Randomized, Double Blind, Pilot Study on the Effect of Intravenous Ibuprofen on Inflammatory Responses in Patients Undergoing Surgery With General Anesthesia: Correlation With Clinical Outcomes
Brief Title: Effect IV Ibuprofen and Inflammatory Responses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012001793
Record Dates: First submitted 2013-05-24; First posted 2013-09-10 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-10

CONDITIONS: Gallbladder Disease
Keywords: laparoscopic cholecystectomy
MeSH Terms: conditions — Gallbladder Diseases | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Active Comparator): 800mg administered IV in 100cc of normal saline over 5 minutes
  Interventions: Drug: ibuprofen
- Sugar water (Placebo Comparator): 100mL of normal saline to be administered over 5 minutes
  Interventions: Other: sugar water/placebo

INTERVENTIONS:
Drug: ibuprofen — single preoperative dose prior to surgery
  Other Names: caldolor
  Arms: Ibuprofen
Other: sugar water/placebo — single preoperative dose prior to surgery
  Other Names: 100mL. intravenous sugar water administered over 5 minutes
  Arms: Sugar water

SUMMARY:
This study is being done because the investigators wish to study ways to improve recovery after surgery. Injury, including surgical injury, causes inflammation. Inflammation is the body's attempt to protect itself and to start the healing process. Some surgical complications are related to the body's natural inflammatory response. Although mainly a healing response, inflammation can also have side effects which delay recovery. The investigators wish to determine the effect of a medication known as ibuprofen on recovery. You may know ibuprofen by the name Advil or Motrin. The medication will be given through the vein prior to the start of the surgery. Three blood samples will be taken, two while the patient is under anesthesia. The subject will be asked to complete several questionnaires.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, two-arm parallel, multi-center study.

Thirty subjects (15 in each arm) will be enrolled. Subjects, over the age of 18, undergoing laparoscopic cholecystectomy under general anesthesia will be screened for eligibility to participate in the study. Subjects will be screened, recruited, and randomized during the preadmission visit or the day of surgery. Eligible subjects will be randomized to one of the two treatment group in a 1:1 ratio to receive either IV ibuprofen or matching placebo. Both men and women will be recruited, and there is no limitation as to racial and ethnic origin.

Participation in the study will not alter the patient's anesthetic management. Routine anesthesia monitors used during general anesthesia will be used. Patients will receive either 800mg IV ibuprofen or placebo pre-operatively. After pre-oxygenation, general anesthesia will be induced with lidocaine (1 mg/kg), propofol (1-2 mg/kg), and fentanyl (up to 5 mcg/kg). Tracheal intubation will be facilitated with rocuronium (0.6 mg/kg). Anesthesia will be maintained with air/oxygen (60%/40%), sevoflurane, and fentanyl. The anesthesiologist will be allowed to administer additional doses of fentanyl at his/her discretion. All patients will receive ondansetron 4 mg prior to the end of operation. Patients will be awakened and extubated in the OR and will be transferred to the Post Anesthesia Care Unit (PACU) after following simple commands. All patients will also be able to receive rescue doses of opioids as indicated by a Numeric Pain Rating Scale score >2 or upon request.

ii. Sample Size Justification: The proposed study is a pilot trial designed to explore the relationship between inflammatory markers and the quality of recovery. To our knowledge this vital connection has never been investigated. Therefore, we cannot use commonly accepted methods of sample size calculations. Mahdy et al examined levels of IL-6, IL-10, and cortisol in patients undergoing urological surgery and treated with indomethacin versus placebo (12). A sample size of twenty three patients per group was sufficient to show a difference in cytokine levels. Tasdogan et al compared levels of interleukin (IL)-1, IL-6, and tumor necrosis factor (TNF)-alpha in patients requiring postoperative ventilation after abdominal surgery and treated with dexmedetomidine versus propofol (18). A sample size of twenty patients per group was sufficient to demonstrate the difference in cytokine concentrations. Kim et al studied changes in cytokine levels in patients undergoing total abdominal hysterectomy and pretreated with clonidine (19). These investigators studied ten patients per group. The sample size was sufficient to demonstrate changes in IL-6 related to surgical stress. Therefore, we believe, that a sample size of 30 patients per group is an adequate sample to demonstrate the changes in level of inflammatory markers and explore the quality of recovery.

iii. IV ibuprofen administration The study drug will be given via intravenous infusion beginning after a placement of the IV line. The dose will be fixed at 800mg infused over 5 minutes.

iv. Inclusion criteria:

1. Adults, 18 and over, who will undergo laparoscopic cholecystectomy.
2. Subject is non-lactating and is either:

   1. Not of childbearing potential
   2. Of childbearing potential but is not pregnant at time of baseline as determined by pre-surgical pregnancy testing.
3. Subject is American Society of Anesthesiologists physical status 1, 2, or 3. v. Exclusion criteria:

1. Cognitively impaired (by history) 2. Subject requires chronic antipsychotic history 3. Subject is anticipated to require an additional surgery within 90 days after the intended surgery 4. Chronic use of steroids or opioids 5. Subject has received treatment with COX inhibitors within 3 days of study entry 6. Subject for whom opiates, benzodiazepines, and COX inhibitors are contraindicated vi. Endpoints: Concentration of the cytokines TNF-alpha, IL-1Beta, IL-2, IL-6, IL-10, and IFN-gamma as well as prostaglandin E2, cortisol and c reactive protein at different time points will be our primary outcome. Changes in mediator levels in the IV ibuprofen versus placebo groups will be compared. Plasma samples will be collected before administration of any drug (after placement of IV lines), before induction, at the end of the surgery in the operating room and 2-3 hours after the end of the surgery in the PACU.

All plasma samples will be analyzed in the laboratory of Susan Gould-Fogerite. The secondary outcome parameters will be the quality of recovery score (QoR-40) to measure quality of recovery from surgery and a simple fatigue scale. Forty questions in five dimensions will be scored by patients on a five-point Likert scale. This assessment was developed and validated by Myles et al (20). Nine points fatigue scale is often used to assess progress of recovery in head trauma patients. Geriatric depression scale and digits backward and forward will be utilized. All metrics will be administered on the day of surgery, before the surgery, 2-3 hours after the end of the surgery in the PACUand on postoperative days 1 and 3. Exploratory analysis will examine whether correlations exist between inflammatory mediator concentrations and the objective measures of recovery and fatigue.

vii. Methods and Procedures

1. Data monitoring plan Adverse events will include events reported by the subject and thought to be associated with the research. Unanticipated problems and adverse events will be gathered by study investigators. Adverse events will be evaluated at each study visit, including follow up telephone calls. Any serious adverse effects will be reported to the Institutional Review Board (IRB) according to regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* undergoing laparoscopic cholecystectomy under general anesthesia
* American Society of Anesthesiologists status of 1, 2 or 3 (as determined by the anesthesiologists)
* not pregnant of breast feeding

Exclusion Criteria:

* cognitively impaired
* using antipsychotic drugs
* chronic use of steroids or opioids
* subject has received COX inhibitors within 3 days if surgery
* subjects for whom opiates, benzodiazepines and COX inhibitors are contraindicated
* subjects with a history of bleeding disorders or peptic ulcer disease

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Bekker, MD, PhD, Principal Investigator — Rutgers/NJMS
Locations (4):
- United States (4):
  - University Hospital, Newark, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - New York University Hospital, New York, New York
  - MT. Sinai Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le V, Kurnutala L, SchianodiCola J, Ahmed K, Yarmush J, Daniel Eloy J, Shapiro M, Haile M, Bekker A. Premedication with Intravenous Ibuprofen Improves Recovery Characteristics and Stress Response in Adults Undergoing Laparoscopic Cholecystectomy: A Randomized Controlled Trial. Pain Med. 2016 Jun;17(6):1163-1173. doi: 10.1093/pm/pnv113. Epub 2016 Feb 18. PMID 26893119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 patients were recruited from the Same Day Surgery Unit at three hospital locations. The dates of recruitment were from 12/1/2011 to 10/2/13.
Pre-assignment Details: Of the 60 patients randomized 5 did not receive study medication. The surgical case was either cancelled or the subjects withdrew consent.
Groups:
- Caldolor/Ibuprofen: 800mg administered IV in 100mL normal saline over 5 minutes prior to surgical incision.
- Placebo: 100mL of normal saline to be administered intravenously over 5 minutes prior to surgical incision.
Period: Overall Study
Arm/Group | Caldolor/Ibuprofen | Placebo
Started | 28 | 27
Plasma Analysis | 24 (complete set of blood samples could not be obtained) | 25 (complete set of blood samples could not be obtained)
Behavior Metrics | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ibuprofen/Caldolor: 800mg administered IV in 100cc of normal saline over 5 minutes
  ibuprofen: single preoperative dose prior to surgery
- Placebo: 100mL of normal saline to be administered over 5 minutes
  sugar water/placebo: single preoperative dose prior to surgery
- Total: Total of all reporting groups
Arm/Group | Ibuprofen/Caldolor | Placebo | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 49
  >=65 years | 5 | 1 | 6
Gender [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 10 | 5 | 15
Region of Enrollment [Number; unit: participants] — All subjects were from the Northeast section of the United States and all were English speaking. The behavioral questionnaires were copyrighted and validated in English only.
  participants
    United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Stress Response Inflammation Markers :Cortisol and C Reactive Protein (CRP)
Description: Serum concentration of cortisol, CRP, drawn in Post Anesthesia Care unit at 2 hours following surgery were compared with those same levels drawn preoperatively and intraoperatively.
Time Frame: 2 hours following end of surgery
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ibuprofen/Caldolor | Placebo
Number analyzed (Participants) | 24 | 25
pg/mL
  cortisol-PACU | 173.6 (29.5) | 289.5 (25.9)
  CRP-PACU | 17 (1) | 17 (1)

2. Post Hoc Outcome: Sympathetic Response: Epinephrine and Norepinephrine Plasma Concentrations
Time Frame: intraoperatively
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ibuprofen/Caldolor | Placebo
Number analyzed (Participants) | 24 | 25
pg/mL
  Epinephrine Intraoperatively | 0.11 (0.03) | 0.23 (0.05)
  Norepinephrine Intraoperatively | 0.52 (0.09) | 1.06 (0.12)

3. Post Hoc Outcome: Immune Response: TNF Alpha
Time Frame: preoperatively-intraoperatively-postoperatively
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Ibuprofen/Caldolor | Placebo
Number analyzed (Participants) | 24 | 25
pg/mL
  TNF a Preop | 12.1 [2.9 to 31.2] | 11.3 [2.9 to 28.1]
  TNFa Intraop | 14 [4.5 to 76.7] | 8.9 [2.8 to 21.0]
  TNF a post op | 11.8 [3.6 to 43.1] | 10.6 [3.6 to 23]

4. Post Hoc Outcome: IL-6
Time Frame: preoperatively-intraoperatively-postoperatively
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Ibuprofen/Caldolor | Placebo
Number analyzed (Participants) | 24 | 25
pg/mL
  IL-6 preoperatively | 1.4 [0.3 to 22.2] | 1.2 [0.4 to 14.5]
  IL-6 intraoperatively | 1.9 [0.4 to 56.4] | 1.1 [0.3 to 22.7]
  IL-6 postoperatively | 8.3 [0.9 to 80.4] | 7.7 [0.5 to 59.1]

5. Secondary Outcome: Immune Response IL-6
Time Frame: 2 hours postoperatively in PACU
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Ibuprofen/Caldolor | Placebo
Number analyzed (Participants) | 24 | 25
pg/mL
  IL-6 PACU | 8.3 [0.9 to 80.4] | 7.7 [0.5 to 59.1]
  IL-6 preoperatively | 1.4 [0.3 to 22.2] | 1.2 [0.4 to 14.5]
  IL-6 intraoperatively | 1.9 [0.4 to 56.4] | 1.1 [0.3 to 22.7]

6. Secondary Outcome: Quality of Recovery-40
Description: Quality of Recovery-40 has been used to assess postoperative recovery from anesthesia where higher score correlate with improved recovery and well being. The survey has 5 domains: comfort scale ranges 1-60 with higher value indicating greater comfort, emotions scale ranges 1-45 with higher value indicating best emotional state, physical independence scale ranges 1-25 with higher value indicating best independence, patient support scale ranges 1-35 with a higher score indicating greater support and pain scale 1-35 with higher number indicating greater relief from pain. Scoring is done for PART A on a scale of 1-5 (1=very poor=none of the time, worst score, 5=excellent=all of the time, best possible score).PART B on a scale of 1-5 (1=very poor or all the time worse score), 5=excellent or none of the time, best score) Perfect score=200.
Time Frame: preoperatively and -postoperative days 1 and 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen/Caldolor | Placebo
Number analyzed (Participants) | 28 | 27
units on a scale
  preop comfort | 56.5 (5.69) | 56.8 (5.12)
  Preop emotion | 42.9 (3.7) | 43 (3.3)
  Preop phy indep | 24.8 (0.7) | 24.6 (1.6)
  preop support | 34.9 (0.19) | 34.5 (1.4)
  preop pain | 34 (1.3) | 33.7 (1.6)
  POD #1 comfort | 58. (2.72) | 51.2 (8.6)
  POD #1 emotion | 44.4 (1.3) | 40.4 (4.1)
  POD #1phy ind | 33.8 (5.7) | 23.5 (3.0)
  POD #1 support | 33.6 (5.7) | 34.2 (3.0)
  POD# 1 pain | 33.6 (1.8) | 27 (7.4)
  POD#3 comfort | 59.4 (0.9) | 55 (4.7)
  POD #3 emotion | 44.8 (0.6) | 43 (2.9)
  POD#3 phy ind | 24.7 (0.8) | 24 (1.6)
  POD#3 support | 34.8 (0.9) | 33.6 (4.2)
  POD#3 pain | 34.5 (0.75) | 30.4 (4.6)

7. Secondary Outcome: Modified Fatigue Severity Scale
Description: This questionnaire contains 9 statements that rate severity of fatigue symptoms. Score 1 indicates strong disagreement with the statement and 7= strong agreement. i.e (I am easily fatigued).Total lowest possible score indicating no fatigue is 9. Total highest possible score is 63 which correlates to severe fatigue, interfering with all activities of daily living.
Time Frame: preoperative-postoperative day 1 and day 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ibuprofen/Caldolor | Placebo
Number analyzed (Participants) | 28 | 27
scores on a scale
  preoperative | 16.7 (8.87) | 16.5 (7.6)
  PACU | 18.6 (11) | 26.9 (14.3)
  Post op day 1 | 15.5 (9.9) | 25 (13.4)
  Post op day #3 | 14.1 (6.57) | 20.8 (8.51)

8. Secondary Outcome: Immune Response:Serum Concentration of IL-10,
Description: .drawn in PACU 2 hours following arrival and compared to preoperative and intraoperative values
Time Frame: 2 hours post arrival in PACU
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Ibuprofen | Sugar Water
Number analyzed (Participants) | 24 | 25
pg/mL
  IL-10 PACU | 8.3 [0.1 to 32.2] | 21.8 [0.1 to 113]
  IL-10 preoperatively | 2.1 [0.0 to 11.2] | 1.3 [0.23 to 24.2]
  IL-10 intraoperatively | 3.3 [0.3 to 76.3] | 2.5 [0.6 to 26.0]
Statistical Analysis 1: Comparison: Ibuprofen vs Sugar Water; Test type: Superiority or Other; p = 0.001, ANOVA

9. Other Pre Specified Outcome: Cytokine Concentrations
Description: IFN y, IL-1B IL-2 were below the limit of detection and no assessments could be made. The lower limit for all cytokine detection was 3.2pg/mL
Time Frame: preoperative-intraoperative-postopoperative
Groups:
- Ibuprofen: 800 mg in 100mL of normal saline over 5 minutes
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Cognitive Recovery.
Description: Digits span forward subject is asked to repeat a series of numbers with increasing number of digits forward. Digit span backward subject is asked to repeat a series of numbers backward with increasing number of digits. Correct response is worth 1 point. Maximum of 14 points for each sub score with a total of 28 points for total score
Time Frame: preoperatively- 2 hours in PACU, Post op day #1, post op day#3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caldolor/Ibuprofen | Placebo
Number analyzed (Participants) | 28 | 27
units on a scale
  preop forward total | 8.4 (1.9) | 8.9 (1.6)
  preoperative forward max len | 6.9 (0.89) | 7.08 (0.8)
  Pre op backward tot | 7.7 (2.08) | 7.7 (1.9)
  Preop backward max len | 5.5 (1.1) | 5.5 (1.1)
  PACU forward tot | 4.7 (2.6) | 4.4 (2.5)
  PACU for max length | 4.8 (1.7) | 4.4 (1.8)
  PACU backward tot | 4.9 (2.9) | 3.1 (2.1)
  PACU back max length | 3.8 (1.7) | 3.0 (1.7)
  Post op #1forward tot | 8.7 (1.6) | 8.8 (1.6)
  Post op day 1max length | 7.03 (0.89) | 7.6 (0.89)
  Post op #1backward tot | 8.2 (1.6) | 7.8 (1.9)
  Post op day #1max length | 5.6 (0.8) | 5.5 (1.2)
  Post op #3 forward tot | 8.7 (1.5) | 8.6 (1.3)
  post #3 for max length | 6.9 (0.89) | 6.8 (0.6)
  post op day #3backward tot | 8.6 (1.8) | 7.6 (1.89)
  post op #3 max length | 6.03 (1.09) | 5.5 (1.2)

11. Secondary Outcome: Geriatric Depression Scale
Description: 15 questions. Score 1 point for each answer selected which indicates depression. Score of 0-5 is normal. A score >5 suggests depression.
Time Frame: Preoperatively, post operative day 1 and post op day3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caldolor/Ibuprofen | Placebo
Number analyzed (Participants) | 28 | 27
units on a scale
  preoperative score | 0.5 (1.1) | 0.7 (1.4)
  PACU | 0.7 (0.9) | 0.9 (0.7)
  post op day #1 | 0.4 (1.1) | 0.4 (0.8)
  post op day #3 | 0.2 (0.8) | 0.12 (0.3)

ADVERSE EVENTS:
Time Frame: -day of surgery to post operative day 3
Arm/Group | Caldolor/Ibuprofen | Placebo
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/27
Other Adverse Events (participants affected / at risk) | 0/28 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caldolor/Ibuprofen (N=28) | Placebo (N=27)
patient unable to be extubated at the end of the surgical procedure (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes